CLINICAL TRIAL: NCT07326527
Title: Effects of a Tele-Based Postural Awareness and Breathing Program on Ergonomic Risk, Sensorimotor Function, and Fatigue in Flute Students: A Randomized Controlled Study
Brief Title: Tele-Based Postural Awareness and Breathing Training for Ergonomic Risk and Fatigue in Flute Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, Assistant Professor, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22.12.2025
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Work-Related Musculoskeletal Risk, Postural Control; Postural Awareness
Keywords: Tele-rehabilitation, Postural Awareness, Ergonomic Risk, Cervical Proprioception, Musicians

STUDY DESIGN:
Intervention Model Description: Study Type: Interventional (Clinical Trial)
  Allocation: Randomized
  Intervention Model: Parallel Assignment
  Masking: None (Open Label)
  Primary Purpose: Prevention
  Number of Arms: 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention / Usual Activity (Active Comparator): Participants do not receive any intervention and continue their usual daily activities and regular flute practice during the 8-week study period.
  Interventions: Other: No Intervention
- Tele-Based Postural Awareness and Pranayama-Based Breathing Program (Experimental): Behavioral: Participants receive an 8-week tele-based program including postural awareness exercises and pranayama-based breathing practices delivered remotely.
  Interventions: Behavioral: Tele-Based Postural Awareness and Pranayama-Based Breathing Program

INTERVENTIONS:
Other: No Intervention — Participants do not receive any intervention and continue their usual daily activities and regular
  Arms: No Intervention / Usual Activity
Behavioral: Tele-Based Postural Awareness and Pranayama-Based Breathing Program — An 8-week tele-rehabilitation program delivered remotely, focusing on postural awareness exercises and pranayama-based breathing practices.
  Arms: Tele-Based Postural Awareness and Pranayama-Based Breathing Program

SUMMARY:
This randomized controlled study investigates the effects of an eight-week tele-based postural awareness and pranayama-based breathing program on work-related ergonomic risk and cervical somatosensory function in flute students. A total of 30 undergraduate flute students were randomly allocated to either an intervention group or a control group.

Participants in the intervention group received a structured tele-rehabilitation program focusing on postural awareness exercises and pranayama-based breathing practices for eight weeks, while the control group did not receive any intervention during the study period.

Primary outcomes include work-related ergonomic risk assessed using the Rapid Upper Limb Assessment (RULA) and cervical somatosensory function evaluated through cervical joint position sense (horizontal, vertical, and global error). Secondary outcomes include deep cervical flexor muscle endurance, perceived fatigue, postural awareness, and musical performance anxiety.

Outcome measures were assessed at baseline and after the eight-week intervention period. The study aims to determine whether a tele-based postural awareness and breathing intervention can effectively reduce ergonomic risk and improve sensorimotor function in flute students who are exposed to prolonged asymmetric postures during instrument practice.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial to examine the effects of a tele-based postural awareness and pranayama-based breathing program on ergonomic risk, cervical somatosensory function, and selected secondary outcomes in flute students.

Thirty undergraduate flute students enrolled in the Faculty of Fine Arts, Department of Music, were recruited and randomly assigned to either an intervention group (n = 15) or a control group (n = 15). Participants were required to have regular flute practice and no history of neurological or musculoskeletal disorders affecting the cervical region.

The intervention group participated in an eight-week tele-rehabilitation program consisting of postural awareness exercises and pranayama-based breathing practices. Sessions were delivered remotely and focused on improving postural alignment, body awareness, controlled breathing, and sensorimotor control relevant to prolonged instrument practice. The control group did not receive any intervention during the study period and continued their usual daily activities.

Outcome assessments were conducted at baseline and at the end of the eight-week intervention period. Primary outcome measures included work-related ergonomic risk, assessed using the Rapid Upper Limb Assessment (RULA), and cervical somatosensory function, evaluated through cervical joint position sense testing in horizontal, vertical, and global directions. Secondary outcome measures included deep cervical flexor muscle endurance, perceived fatigue assessed using the Modified Borg Scale, postural awareness, and musical performance anxiety assessed using a validated questionnaire.

This study aims to evaluate the feasibility and effectiveness of a tele-based postural awareness and breathing intervention in reducing ergonomic risk and improving sensorimotor function in flute students exposed to prolonged asymmetric postures during musical practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 28 years
* Enrolled as a student in the Department of Music at the Faculty of Fine Arts or Faculty of Education
* Has been playing the flute for at least 3 years
* Willing to participate in the study and able to provide informed consent

Exclusion Criteria:

* History of upper extremity surgery
* Presence of any diagnosed neurological disorder
* History of cardiovascular disease
* Presence of an acute musculoskeletal injury that could affect performance

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Total RULA Score and RULA B Score | Baseline and 8 weeks
  Postural ergonomic risk is assessed during flute performance using the Rapid Upper Limb Assessment (RULA), which evaluates neck, trunk, and upper limb posture. The total RULA score ranges from 1 to 7, with higher scores indicating greater ergonomic risk.
Cervical Somatosensory Function (Joint Position Sense - JPS) | Baseline and 8 weeks
  Cervical joint position sense is assessed using a laser-pointer repositioning method during flexion, extension, and rotation movements. Horizontal, vertical, and global angular errors are calculated. Higher error values indicate reduced proprioceptive accuracy.

SECONDARY OUTCOMES:
Postural Habits and Awareness Scale (PAFÖ) total score | Baseline and 8 weeks
  A self-reported scale assessing postural habits and postural awareness across four domains: posture habit and awareness, awareness of posture-disturbing factors, position awareness, and ergonomic awareness. Higher scores indicate better postural awareness.
Deep Cervical Flexor Muscle Endurance | Baseline and 8 weeks
  Participants maintain a chin-tuck with slight head lift in supine position. The duration the position is maintained without compensation is recorded in seconds.
Modified Borg Scale score | Baseline and 8 weeks
  Fatigue is assessed using the Modified Borg Scale, which measures perceived exertion and fatigue following classes, rehearsals, and performances.
Kenny Music Performance Anxiety Inventory (K-MPAI) total score | Baseline and 8 weeks
  A validated 25-item questionnaire assessing musical performance anxiety across psychological, somatic, and control-related domains. Higher scores indicate greater performance anxiety.Total score on the Kenny Music Performance Anxiety Inventory (range 0-240), where higher scores indicate greater performance anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Alaaddin Keykubat University, Alanya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves small sample sizes and includes sensitive personal, performance, and health-related information. Data sharing could increase the risk of participant identification. In accordance with the approval of the institutional ethics committee and applicable data protection regulations, the data will be used only by the research team for the purposes of this study.